CLINICAL TRIAL: NCT01415778
Title: Bioequivalence Study of ICI176,334-1 in Japanese Healthy Male Subjects - Evaluation of Bioequivalence of ICI176,334-1 and Casodex 80 mg Tablet -
Brief Title: Bioequivalence of ICI176,334-1 in Japanese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D6874L00025
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Bioequivalence; pharmacokinetics; safety; bicalutamide; Casodex; Japanese; healthy subject
MeSH Terms: interventions — bicalutamide; Tablets

ARMS (4):
- Active 1 (Experimental): 12 subjects will receive ICI176,334-1 and Casodex 80 mg tablet
  Interventions: Drug: ICI176,334-1; Drug: Casodex 80 mg tablet
- Active 2 (Experimental): 12 subjects will receive ICI176,334-1 and Casodex 80 mg tablet
  Interventions: Drug: ICI176,334-1; Drug: Casodex 80 mg tablet
- Active 3 (Experimental): 12 subjects will receive ICI176,334-1 and Casodex 80 mg tablet
  Interventions: Drug: ICI176,334-1; Drug: Casodex 80 mg tablet
- Active 4 (Experimental): 12 subjects will receive ICI176,334-1 and Casodex 80 mg tablet
  Interventions: Drug: ICI176,334-1; Drug: Casodex 80 mg tablet

INTERVENTIONS:
Drug: ICI176,334-1 — Subject will receive single dose of ICI176,334-1
Drug: Casodex 80 mg tablet — Subject will receive single dose of Casodex 80 mg tablet

SUMMARY:
The purpose of this study is to investigate the bioequivalence of ICI176,334-1 in Japanese healthy male subjects.

DETAILED DESCRIPTION:
Bioequivalence study of ICI176,334-1 in Japanese healthy male subjects - evaluation of bioequivalence of ICI176,334-1 and Casodex 80 mg tablet -

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Japanese healthy male subjects aged 20 to 45 years
* Male subjects should be willing to use barrier contraception ie, condoms, until 3 months after the last dose of investigational product
* Have a body mass index (BMI) between 17 and 27 kg/m2
* Eligible based on the physical findings, supine BP, pulse rate, ECG and laboratory assessments, as judged by the investigator(s)

Exclusion Criteria:

* Presence of any disease under medical treatment
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunological, blood, endocrine, neurological or mental disease to interfere with absorption, distribution, metabolism or excretion of drugs judged by investigator(s)
* Presence of any infectious disease, such as bacteria, virus and fungus
* Presence of allergic disorder, such as asthma, pollen disease or atopic dermatitis, and judged as necessary any medical treatment
* Any large surgical history of gastrointestinal tract such as gastric/intestinal resection or suturation

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To investigate the bioequivalence of ICI176,334-1 by assessment of maximum plasma concentration (Cmax) | Blood samples are taken repeatedly for 72 hours and also taken occasionally up to 672 hours after each dose period
To investigate the bioequivalence of ICI176,334-1 by assessment of time to Cmax (tmax) | Blood samples are taken repeatedly for 72 hours and also taken occasionally up to 672 hours after each dose period
To investigate the bioequivalence of ICI176,334-1 by assessment of area under the plasma concentration curve (AUC) | Blood samples are taken repeatedly for 72 hours and also taken occasionally up to 672 hours after each dose period
To investigate the bioequivalence of ICI176,334-1 by assessment of t1/2 of bicalutamide | Blood samples are taken repeatedly for 72 hours and also taken occasionally up to 672 hours after each dose period

SECONDARY OUTCOMES:
To assess the safety by assessment of adverse event | Screening day up to 35 to 42 days (follow-up)
To assess the safety by assessment of vital signs | Collect prior to treatment and up to 35 to 42 days (follow-up) after the last dose.
To assess the safety by assessment of electrocardiograms (ECGs) | Collect prior to treatment and up to 35 to 42 days (follow-up) after the last dose.